CLINICAL TRIAL: NCT03282188
Title: A Clinical Study to Evaluate the Biological Effects of Intravenous Wild-type Reovirus (Reolysin®), With of Without GM-CSF, in Advanced Melanoma
Brief Title: REO13 Melanoma With of Without GM-CSF
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn by Sponsor
Sponsor: University of Leeds (Other)
Collaborators: Yorkshire Cancer Research (Other)
Responsible Party: Principal Investigator, Christy Ralph, Associate Professor and Medical Oncology Consultant, University of Leeds
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: MO15/121
Record Dates: First submitted 2017-08-30; First posted 2017-09-13 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Melanoma; Cancer of Skin
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — reolysin; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Intervention Model Description: This is a open-label, non-randomised, single centre study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GROUP A (Reovirus only) (Experimental): Group A patients will receive an initial low 'immunisation' dose of intravenous reovirus (1x108 TCID50), to ensure that neutralising antibody (NAB) levels have risen by the time a full cycle of reovirus is given. Group A patients will then receive only 1 cycle of treatment which will comprise of reovirus only at 1x1010 TCID50 as a 1-hour IV infusion on 2 consecutive days.
  Interventions: Biological: Reolysin
- GROUP B (Reovirus plus GM-CSF) (Experimental): Group B patients will receive an initial low 'immunisation' dose of intravenous reovirus (1x108 TCID50), to ensure that neutralising antibody (NAB) levels have risen by the time a full cycle of reovirus plus GM-CSF is given. Group B patients will be given a subcutaneous injection of GM-CSF (50mcg/day) for 3 days, followed by only 1 cycle of treatment which will comprise of reovirus at 1x1010 TCID50 as a 1-hour IV infusion on 2 consecutive days
  Interventions: Biological: Reolysin; Drug: GM-CSF

INTERVENTIONS:
Biological: Reolysin — Reolysin® is a proprietary isolate of Reovirus Type 3 Dearing, a non-enveloped human reovirus with a genome that consists of 10 segments of double-stranded RNA. The human reovirus possesses an innate ability to replicate specifically in transformed cells possessing an activated Ras signalling pathway, a situation often found in malignant cells. Reovirus has been shown to reach and target melanoma cancer cells.
Drug: GM-CSF — GM-CSF is a recombinant human granulocyte-macrophage colony stimulating factor (rhu GM-CSF) produced by recombinant DNA technology in a yeast (S. cerevisiae) expression system. GM-CSF is a hematopoietic growth factor which stimulates proliferation and differentiation of hematopoietic progenitor cells. GM-CSF is a key cytokine in the differentiation of dendritic cells. It has been used as an immune adjuvant in therapeutic vaccines in pre-clinical and clinical studies, administered as cytokine released from gene-transduced tumour or stromal cells or as recombinant protein. At low doses GM-CSF may enhance migration and differentiation of dendritic cells to local antigen presentation, and is a potent adjuvant to generate specific systemic anti-tumour efficacy.
  Other Names: LEUKINE; Sargramostim
  Arms: GROUP B (Reovirus plus GM-CSF)

SUMMARY:
Open-label, non-randomised, single centre study which will assess the presence of reovirus (Reolysin®), following intravenous administration with or without Granulocyte-macrophage colony-stimulating factor (GM-CSF) given to patients prior to surgery for metastatic melanoma. All patients will receive an initial low 'immunisation' dose of intravenous reovirus. Patients will be enrolled sequentially in to each of the two cohorts receiving either reovirus alone, or reovirus plus GM-CSF. For this study we anticipate 8-16 evaluable patients, up to 8 for each group. The endpoints of this study will compare the 2 treatment groups for reovirus tumour infiltration and replication. Compare the neutralising antibody development and cell-mediated immune response and identify any adverse events and laboratory toxicities.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, single centre study of intravenous reovirus (Reolysin®) with or without Granulocyte-macrophage colony-stimulating factor (GM-CSF) given to patients prior to surgery for metastatic melanoma. Patients will be eligible if undergoing surgery for local control of lymph node involvement (with or without stage 4 metastases) or if planned for resection of cutaneous, subcutaneous, musculoskeletal or visceral metastases for local control, palliation of symptoms or personal choice.

All patients will receive an initial low 'immunisation' dose of intravenous reovirus (1x108 TCID50), to ensure that neutralising antibody (NAB) levels have risen by the time a full cycle of reovirus +/- GM-CSF is given. All patients will receive only 1 cycle of treatment which will comprise: i) For reovirus alone patients (Group A), 1x1010 TCID50 as a 1-hour IV infusion on 2 consecutive days; ii) For reovirus plus GM-CSF patients (Group B), subcutaneous GM-CSF (50mcg/day) for 3 days, followed by 2 days of reovirus. Both doses of reovirus will be at 1x1010 TCID50.

Patients will be enrolled sequentially into each of the two cohorts receiving intravenous reovirus alone, or reovirus plus GM-CSF. The addition of GM-CSF is designed to address effects on the translational objectives/endpoints of this study, rather than primary toxicity, although all patients will be monitored for safety. Clinical assessment will be performed at screening (within 14 days of start of treatment), at day 1 (1st GM-CSF dose/none), day 8 and at the final study visit (40 days (+/- 14 days) post treatment with reovirus). Safety bloods will be taken at screening, at treatment (Day 1), before each dose of reovirus (Day 4 & 5), at Day 8 and at the final study visit (Day 40). Immunological assays, including reovirus antibody levels, will be performed before low-dose reovirus priming (Day -10 to -6), pre-treatment on Day 1, on Day 4 and 5 (pre-reovirus infusion and 60 minutes post-infusion), Day 8, and at the final study visit (Day 40). Patients with accessible skin or subcutaneous metastases will be asked for an optional additional pre-treatment biopsy which will be taken before low-dose reovirus priming.

All procedures will be performed as an outpatient or day case, apart from surgery in melanoma patients requiring admission as part of standard clinical care. Imaging will be as for standard clinical care only. Following surgical resection the tumour will be assessed for viral status and anti-tumour effects by e.g. standard histology, immunohistochemistry, RT-PCR and electron microscopy. Further imaging and follow-up beyond the final study visit (Day 40 +/- 14 days) will be as for standard clinical care only.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female subjects with histologically diagnosed melanoma.
2. Be at least 18 years of age.
3. Be appropriate for resection of advanced melanoma (Stage 3/4). Patients may or may not have more widespread metastatic disease.
4. Have completed any previous systemic chemotherapy, radiotherapy or surgery (except biopsies) at least 28 days before entry into the study.
5. Have NO continuing acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures, i.e., all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0) Grade ≤1.
6. Have an ECOG Performance Score of 0 or 1.
7. Have a life expectancy of at least 3 months.
8. Have baseline laboratory results at the time of consent as follows:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109 [SI units 109/L]
   2. Platelets ≥ 100 x109 [SI units 109/L] (without platelet transfusion)
   3. Haemoglobin ≥ 9.0 g/dL [SI units gm/L] (with or without RBC transfusion)
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
   5. Bilirubin ≤ 1.5 x ULN
   6. AST/ALT ≤ 2.5 x ULN
   7. Negative serum pregnancy test for females of childbearing potential.
9. Have signed informed consent.
10. Be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests

Exclusion Criteria:

1. Be on concurrent therapy with any other investigational anticancer agent while on study.
2. Be on immunosuppressive therapy other than steroids.
3. Have known HIV infection or hepatitis B or C.
4. Be pregnant or breast feeding. Female patients must agree to use effective contraception, be surgically sterile, or be postmenopausal. Male patients must agree to use effective contraception or be surgically sterile.
5. Have clinically significant cardiac disease (New York Heart Association, Class III or IV) including clinically significant arrhythmia, uncontrolled angina pectoris, or myocardial infarction within 1 year prior to study entry.
6. Have dementia or altered mental status that would prohibit informed consent.
7. Have any other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Comparison between treatment groups of reovirus tumour infiltration by immunohistochemistry (IHC) | Through study completion, an average of 18 months

SECONDARY OUTCOMES:
Comparison between treatment groups of reovirus tumour replication, as assessed by qRT-PCR | Through study completion, an average of 18 months
Comparison between treatment groups of neutralising antibody development development and cell-mediated immune response | Through study completion, an average of 18 months
Comparison between treatment groups of cell-mediated immune response | Through study completion, an average of 18 months